CLINICAL TRIAL: NCT02713347
Title: Palliative Care to Improve Quality of Life in CHF and COPD
Brief Title: Advancing Symptom Alleviation With Palliative Treatment
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: IIR 14-346
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Heart Failure; Pulmonary Disease, Chronic Obstructive; Emphysema; Pulmonary Fibrosis, Interstitial Lung Disease
Keywords: Quality of Life; Symptom Assessment; Palliative Care; Disease Management; Delivery of Health Care; Advance Care Planning
MeSH Terms: conditions — Heart Failure; Pulmonary Disease, Chronic Obstructive; Emphysema; Pulmonary Fibrosis; Lung Diseases, Interstitial

STUDY DESIGN:
Intervention Model Description: Parallel
Who Masked: Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ADAPT Intervention (Experimental): The intervention includes 3 components:
  1. nurse (RN) follows structured algorithms to help patients with symptoms, specifically breathlessness, fatigue, and pain.
  2. social worker provides structured counseling targeting adjustment to illness and depression and advance care planning.
  3. collaborative care model of care delivery, in which the nurse and social worker meet weekly with a primary care provider and palliative care specialist. This team makes medical recommendations to the intervention subjects' providers and supervises the nurse and social worker. The team has as-needed consultation with a cardiologist or pulmonologist.
  The nurse and social worker visits are in-person or by phone.
  Interventions: Behavioral: ADAPT Intervention
- Enhanced usual care (No Intervention): Patients in the control group will continue to receive care at the discretion of their providers, which may include referrals to and ongoing care from cardiology, pulmonary, palliative care, or mental health. They will also have the same amount of interaction with research assistants as the intervention patients, completing questionnaires and participating in study visits at the same frequency. Patients' providers will be given the results of baseline depression surveys if they screen positive for depression, and patients will be given an information sheet that outlines self-care for CHF or COPD.

INTERVENTIONS:
Behavioral: ADAPT Intervention — The intervention includes 3 components:
  1. nurse (RN) follows structured algorithms to help patients with symptoms, specifically breathlessness, fatigue, and pain.
  2. social worker provides structured counseling targeting adjustment to illness and depression and advance care planning.
  3. collaborative care model of care delivery, in which the nurse and social worker meet weekly with a primary care provider and palliative care specialist. This team makes medical recommendations to the intervention subjects' providers and supervises the nurse and social worker. The team has as-needed consultation with a cardiologist or pulmonologist. The nurse and social worker visits are in-person or by phone.
  Arms: ADAPT Intervention

SUMMARY:
Chronic heart failure (CHF), chronic obstructive pulmonary disease (COPD), and interstitial lung disease (i.e., pulmonary fibrosis) are common serious illnesses. Despite disease-specific medical care, people with these illnesses often left with poor quality of life (i.e., burdensome symptoms, impaired function). Furthermore, while these illnesses are leading causes of hospitalization and mortality, few people with these illnesses engage in advance care planning, the process of considering and communicating healthcare values and goals. The investigators are conducting a randomized clinical trial to study a symptom management, psychosocial care and advance care planning intervention to improve quality of life. The study is important because it aims to improve quality of life and provision of care according to peoples' goals and preferences in common, burdensome illnesses. Furthermore, this study will generate information that supports the broader dissemination and implementation of the intervention and informs the development of future palliative care and team-based interventions in the VA.

DETAILED DESCRIPTION:
Chronic heart failure (CHF), chronic obstructive pulmonary disease (COPD) and interstitial lung disease (i.e., pulmonary fibrosis) have commonalities that make them ideal for early palliative care provided alongside disease-specific treatments. Quality of life is reduced in these illnesses because, despite disease-specific treatments, the same symptoms (e.g., shortness of breath, fatigue) often persist in these illnesses. Quality of life is also reduced because between 50-60% of people with either illness have clinically significant depressive symptoms. Finally, while CHF, COPD, and interstitial lung disease are leading causes of hospitalization and mortality, few people with these illnesses engage in advance care planning. Providing palliative care concomitantly with other medical care offers an important opportunity to improve quality of life and advance care planning for people with CHF, COPD, or interstitial lung disease. For other conditions such as lung cancer, when provided early, prior to the end of life, palliative care improves quality of life, depressive symptoms, and survival while reducing health care utilization. While palliative care has been well-studied in patients with advanced cancer, it has not been adequately studied in CHF, COPD, or interstitial lung disease. The goal of this project is to determine whether the benefits of early palliative care extend to CHF, COPD or interstitial lung disease.

The investigators developed and demonstrated early success with a patient-centered palliative care intervention to improve quality of life (i.e., symptoms, function) and advance care planning in CHF and COPD. The intervention consists of the following components: (1) algorithm-guided management of breathlessness, fatigue, and pain, provided by a nurse; the algorithms supplement disease-focused treatments with palliative and behavioral treatments; (2) a 6-session psychosocial care program targeting adjustment to illness and depression, provided by a social worker; and (3) engagement of patients and providers in advance care planning. The nurse and social worker are teamed with a palliative care specialist and representative primary care provider in brief weekly meetings. The team is integrated into primary care through nurse interaction with primary care providers and through electronic medical record communication.

The investigators will conduct a hybrid effectiveness and implementation study. Population-based sampling methods will be used to enroll 300 Veterans with CHF, COPD, or interstitial lung disease who have poor quality of life and are at high risk for hospitalization or death. The primary aim is to test the effectiveness of the intervention in a randomized controlled trial (intervention vs. enhanced usual care) in two VA health care systems. In a secondary aim, the investigators will examine the implementation of the intervention to guide future implementation and dissemination, increase the relevance to operational partners, and maximize the effectiveness of subsequent palliative care and team-based interventions.

Aim 1: Determine the effect of the intervention on (a) quality of life as a primary outcome, and (b) depression, symptom burden, advance care planning communication and documentation, disease-specific health status, emergency department visits, hospitalizations, and mortality as secondary outcomes.

Aim 2: Examine the implementation of the intervention.

Aim 2a: Assess the degree, barriers, and facilitators of implementation of various components. Identify which intervention components and processes are most critical from the perspectives of patients, intervention team members, and primary care providers whose patients received the intervention.

Aim 2b. Evaluate the resources (e.g., personnel time and other costs) associated with the intervention, and estimate the resources needed for implementation and maintenance in other VA settings.

The proposed study is significant because it addresses patient-centered needs in illnesses that are major sources of disability. The study is innovative because it tests the effectiveness of palliative care in CHF, COPD, and interstitial lung disease, leading causes of death among Veterans. In addition, the intervention is integrated into primary care, and the intervention components are structured to ease replication, implementation, and dissemination.

ELIGIBILITY:
Inclusion Criteria:

* Veterans enrolled in VA Eastern Colorado Health Care System or VA Puget - Sound Health Care System
* Diagnosis of CHF, pulmonary fibrosis, or COPD in 2 years prior to enrollment
* High risk for hospitalization and death
* Poor quality of life
* Symptomatic
* Primary care or other provider who is willing to facilitate intervention medical recommendations
* Able to read and understand English
* Consistent access to and able to use a standard telephone

Exclusion Criteria:

* Previous diagnosis of dementia
* Active substance abuse
* Comorbid metastatic cancer
* Nursing home resident
* Heart or lung transplant or left ventricular assist device (LVAD)
* Currently receiving hospice, palliative or home-based primary care
* Currently pregnant
* Currently a prisoner

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Bekelman, MD MPH, Principal Investigator — Rocky Mountain Regional VA Medical Center, Aurora, CO
Locations (2):
- United States (2):
  - Rocky Mountain Regional VA Medical Center, Aurora, CO, Aurora, Colorado
  - VA Puget Sound Health Care System Seattle Division, Seattle, WA, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
We will consider a plan to share individual patient data in consultation with VA privacy, information security, and research and development offices.

REFERENCES:
- [Background] Bekelman DB, Johnson-Koenke R, Ahluwalia SC, Walling AM, Peterson J, Sudore RL. Development and Feasibility of a Structured Goals of Care Communication Guide. J Palliat Med. 2017 Sep;20(9):1004-1012. doi: 10.1089/jpm.2016.0383. Epub 2017 Apr 19. PMID 28422561
- [Background] Kavalieratos D, Gelfman LP, Tycon LE, Riegel B, Bekelman DB, Ikejiani DZ, Goldstein N, Kimmel SE, Bakitas MA, Arnold RM. Palliative Care in Heart Failure: Rationale, Evidence, and Future Priorities. J Am Coll Cardiol. 2017 Oct 10;70(15):1919-1930. doi: 10.1016/j.jacc.2017.08.036. PMID 28982506
- [Background] Bekelman DB, Johnson-Koenke R, Bowles DW, Fischer SM. Improving Early Palliative Care with a Scalable, Stepped Peer Navigator and Social Work Intervention: A Single-Arm Clinical Trial. J Palliat Med. 2018 Jul;21(7):1011-1016. doi: 10.1089/jpm.2017.0424. Epub 2018 Feb 20. PMID 29461908
- [Background] Bekelman DB, Allen LA, McBryde CF, Hattler B, Fairclough DL, Havranek EP, Turvey C, Meek PM. Effect of a Collaborative Care Intervention vs Usual Care on Health Status of Patients With Chronic Heart Failure: The CASA Randomized Clinical Trial. JAMA Intern Med. 2018 Apr 1;178(4):511-519. doi: 10.1001/jamainternmed.2017.8667. PMID 29482218
- [Background] Portz JD, Cognetta S, Bekelman DB. Potential Technology Development for Palliative Care. J Palliat Med. 2018 Jul;21(7):899-900. doi: 10.1089/jpm.2018.0126. No abstract available. PMID 29975619
- [Background] Bekelman DB, Knoepke CE, Turvey C. Identifying critical psychotherapy targets in serious cardiac conditions: The importance of addressing coping with symptoms, healthcare navigation, and social support. Palliat Support Care. 2019 Oct;17(5):531-535. doi: 10.1017/S1478951518001037. PMID 30702055
- [Background] Graney BA, Au DH, Baron AE, Cheng A, Combs SA, Glorioso TJ, Paden G, Parsons EC, Rabin BA, Ritzwoller DP, Stonecipher JJ, Turvey C, Welsh CH, Bekelman DB. Advancing Symptom Alleviation with Palliative Treatment (ADAPT) trial to improve quality of life: a study protocol for a randomized clinical trial. Trials. 2019 Jun 13;20(1):355. doi: 10.1186/s13063-019-3417-1. PMID 31196156
- [Background] Bekelman DB. Improving Primary and Specialist Palliative Care in Cardiovascular Disease. JAMA Netw Open. 2019 May 3;2(5):e192356. doi: 10.1001/jamanetworkopen.2019.2356. No abstract available. PMID 31050771
- [Background] Portz JD, Fruhauf C, Bull S, Boxer RS, Bekelman DB, Casillas A, Gleason K, Bayliss EA. "Call a Teenager... That's What I Do!" - Grandchildren Help Older Adults Use New Technologies: Qualitative Study. JMIR Aging. 2019 Jun 6;2(1):e13713. doi: 10.2196/13713. PMID 31518274
- [Background] Portz JD, Bayliss EA, Bull S, Boxer RS, Bekelman DB, Gleason K, Czaja S. Using the Technology Acceptance Model to Explore User Experience, Intent to Use, and Use Behavior of a Patient Portal Among Older Adults With Multiple Chronic Conditions: Descriptive Qualitative Study. J Med Internet Res. 2019 Apr 8;21(4):e11604. doi: 10.2196/11604. PMID 30958272
- [Background] Buck HG, Bekelman D, Cameron J, Chung M, Hooker S, Pucciarelli G, Stromberg A, Riegel B, Vellone E. A body of work, a missed opportunity: Dyadic research in older adults. J Am Geriatr Soc. 2019 Apr;67(4):854-855. doi: 10.1111/jgs.15749. Epub 2019 Jan 11. No abstract available. PMID 30632603
- [Background] Giannitrapani KF, Walling AM, Garcia A, Foglia M, Lowery JS, Lo N, Bekelman D, Brown-Johnson C, Haverfield M, Festa N, Shreve ST, Gale RC, Lehmann LS, Lorenz KA. Pilot of the Life-Sustaining Treatment Decisions Initiative Among Veterans With Serious Illness. Am J Hosp Palliat Care. 2021 Jan;38(1):68-76. doi: 10.1177/1049909120923595. Epub 2020 May 8. PMID 32383388
- [Background] Brown-Johnson C, Haverfield MC, Giannitrapani KF, Lo N, Lowery JS, Foglia MB, Walling AM, Bekelman DB, Shreve ST, Lehmann LS, Lorenz KA. Implementing Goals-of-Care Conversations: Lessons From High- and Low-Performing Sites From a VA National Initiative. J Pain Symptom Manage. 2021 Feb;61(2):262-269. doi: 10.1016/j.jpainsymman.2020.07.040. Epub 2020 Aug 8. PMID 32781166
- [Background] Hadler RA, Curtis BR, Ikejiani DZ, Bekelman DB, Harinstein M, Bakitas MA, Hess R, Arnold RM, Kavalieratos D. "I'd Have to Basically Be on My Deathbed": Heart Failure Patients' Perceptions of and Preferences for Palliative Care. J Palliat Med. 2020 Jul;23(7):915-921. doi: 10.1089/jpm.2019.0451. Epub 2020 Jan 9. PMID 31916910
- [Background] Schenker Y, Ellington L, Bell L, Kross EK, Rosenberg AR, Kutner JS, Bickel KE, Ritchie C, Kavalieratos D, Bekelman DB, Mooney KB, Fischer SM. The National Postdoctoral Palliative Care Research Training Collaborative: History, Activities, Challenges, and Future Goals. J Palliat Med. 2021 Apr;24(4):545-553. doi: 10.1089/jpm.2020.0411. Epub 2020 Sep 21. PMID 32955969
- [Background] Cooney TM, Proulx CM, Bekelman DB. Changes in Social Support and Relational Mutuality as Moderators in the Association Between Heart Failure Patient Functioning and Caregiver Burden. J Cardiovasc Nurs. 2021 May-Jun 01;36(3):212-220. doi: 10.1097/JCN.0000000000000726. PMID 32740225
- [Background] Deng LR, Masters KS, Schmiege SJ, Hess E, Bekelman DB. Two Factor Structures Possible for the FACIT-Sp in Patients With Heart Failure. J Pain Symptom Manage. 2021 Nov;62(5):1034-1040. doi: 10.1016/j.jpainsymman.2021.05.009. Epub 2021 May 19. PMID 34019976
- [Background] Deng LR, Masters KS, Schmiege SJ, Hess E, Bekelman DB. Factor Structure of Functional Assessment of Chronic Illness Therapy: Spiritual Well-Being Scale in Patients with Heart Failure Depends on Method Used. J Palliat Med. 2021 Jun;24(6):807-808. doi: 10.1089/jpm.2021.0064. No abstract available. PMID 34061665
- [Background] Ma JE, Haverfield M, Lorenz KA, Bekelman DB, Brown-Johnson C, Lo N, Foglia MB, Lowery JS, Walling AM, Giannitrapani KF. Exploring expanded interdisciplinary roles in goals of care conversations in a national goals of care initiative: A qualitative approach. Palliat Med. 2021 Sep;35(8):1542-1552. doi: 10.1177/02692163211020473. Epub 2021 Jun 3. PMID 34080488
- [Background] Portz JD, Graney BA, Bekelman DB. "Made Me Realize That Life Is Worth Living": A Qualitative Study of Patient Perceptions of a Primary Palliative Care Intervention. J Palliat Med. 2022 Jan;25(1):28-38. doi: 10.1089/jpm.2021.0015. Epub 2021 Jul 14. PMID 34264752
- [Result] Bekelman DB, Feser W, Morgan B, Welsh CH, Parsons EC, Paden G, Baron A, Hattler B, McBryde C, Cheng A, Lange AV, Au DH. Nurse and Social Worker Palliative Telecare Team and Quality of Life in Patients With COPD, Heart Failure, or Interstitial Lung Disease: The ADAPT Randomized Clinical Trial. JAMA. 2024 Jan 16;331(3):212-223. doi: 10.1001/jama.2023.24035. PMID 38227034
- [Derived] Ladebue A, Barnard JG, Haverhals LM, Morgan B, Blanchard K, Sloan M, Bekelman DB. Advancing Symptom Alleviation With Palliative Treatment (ADAPT): A Qualitative Study to Understand How a Nurse and Social Worker Palliative Telecare Team Improved Quality of Life in Chronic Illness. J Appl Gerontol. 2025 May 22:7334648251343506. doi: 10.1177/07334648251343506. Online ahead of print. PMID 40400366
- [Derived] Lange AV, Feser WJ, Hess E, Baron AE, Ma JE, Bekelman DB. Serious Illness Communication in a Randomized Trial of a Nurse and Social Worker Palliative Telecare Team. J Am Geriatr Soc. 2025 Mar 22. doi: 10.1111/jgs.19445. Online ahead of print. PMID 40119839

RESULTS

PARTICIPANT FLOW:
Groups:
- ADAPT Intervention: The intervention includes 3 components:
  1. nurse (RN) follows structured algorithms to help patients with symptoms, specifically breathlessness, fatigue, and pain.
  2. social worker provides structured counseling targeting adjustment to illness and depression and advance care planning.
  3. collaborative care model of care delivery, in which the nurse and social worker meet weekly with a primary care provider and palliative care specialist. This team makes medical recommendations to the intervention subjects' providers and supervises the nurse and social worker. The team has as-needed consultation with a cardiologist or pulmonologist.
  The nurse and social worker visits are in-person or by phone.
  ADAPT Intervention: The intervention includes 3 components:
  1. nurse (RN) follows structured algorithms to help patients with symptoms, specifically breathlessness, fatigue, and pain.
  2. social worker provides structured counseling targeting adjustment to illness and depression and advance care planning.
  3. collaborative care model of care delivery, in which the nurse and social worker meet weekly with a primary care provider and palliative care specialist. This team makes medical recommendations to the intervention subjects' providers and supervises the nurse and social worker. The team has as-needed consultation with a cardiologist or pulmonologist. The nurse and social worker visits are in-person or by phone.
Period: Baseline to 4 Months
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Started | 154 | 152
Completed | 120 | 129
Not Completed | 34 | 23
Period: 4 Months to 6 Months
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Started (The number eligible for follow-up at this time period was entered. The investigators allowed patients to miss a study time point and be eligible to complete surveys at subsequent time points. Participants who withdrew or deceased were not eligible for follow-up.) | 148 | 148
Completed | 122 | 122
Not Completed | 26 | 26
Period: 6 Months to 12 Months
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Started (The number eligible for follow-up at this time period was entered. We allowed patients to miss a study time point and be eligible to complete surveys at subsequent time points. Participants who withdrew or deceased were not eligible for follow-up.) | 146 | 143
Completed | 107 | 111
Not Completed | 39 | 32

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ADAPT Intervention | Enhanced Usual Care | Total
Number analyzed (Participants) | 154 | 152 | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 34 | 82
  >=65 years | 106 | 118 | 224
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (8.0) | 68.9 (7.4) | 68.9 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 15 | 30
  Male | 139 | 137 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 128 | 127 | 255
  Unknown or Not Reported | 16 | 17 | 33
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 13 | 7 | 20
  White | 118 | 127 | 245
  More than one race | 16 | 14 | 30
  Unknown or Not Reported | 3 | 0 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 154 | 152 | 306

OUTCOME MEASURES:

1. Primary Outcome: Function Assessment of Chronic Illness Therapy-General (FACT-G)
Description: The FACT-G is a widely used, valid, reliable, and responsive self-report measure of health-related quality of life that includes domains of physical, social/family, emotional, and functional well-being. The primary outcome will be the difference in FACT-G score at 6 months. The total score range is 0-108 with a higher score meaning greater quality of life.
Time Frame: 6 months
Population: Total number reported here may be inconsistent from the participant flow number because (1) participants could skip completion of a survey and maintain enrollment in the study, and (2) FACT-G surveys may not have been completed enough for analysis (i.e., there were too many missing FACT-G items to score the measure).
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 153 | 147
score on a scale | 59.0 (4.0) | 54.0 (4.0)

2. Secondary Outcome: General Symptom Distress Scale (GSDS)
Description: The General Symptom Distress Scale (GSDS) is a single item measure of overall symptom distress that is reliable and valid and asks, "In general, how distressing are all of your symptoms to you?" Minimum value 0 Maximum value 10 Higher scores mean more distress
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 153 | 150
score on a scale | 5.56 (0.64) | 6.0 (0.64)

3. Secondary Outcome: Patient Health Questionnaire-8 (PHQ-8)
Description: The PHQ-8 is a 8-item valid and reliable instrument that provides a continuous measure of depressive symptoms and is 88% sensitive and specific for a diagnosis of major depressive disorder. The PHQ-8 was developed in medically-ill outpatients. Score range 0-24 points with a higher score indicating more depressive symptoms.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 154 | 152
score on a scale | 10.02 (1.43) | 11.58 (1.42)

4. Secondary Outcome: Kansas City Cardiomyopathy Questionnaire- Short Form (KCCQ-SF)
Description: The KCCQ-SF is a self-administered questionnaire that measures heart failure-specific health status. The KCCQ-SF is reliable, sensitive to clinical change, and predicts hospitalization and mortality. The KCCQ-SF will be administered to participants with heart failure. Score range 0-100 and higher scores indicate better health status.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 51 | 50
score on a scale | 47.6 (3.47) | 43.05 (3.52)

5. Secondary Outcome: Clinical COPD Questionnaire (CCQ)
Description: The CCQ is a self-administered 10-item measure of COPD symptoms, functioning, and emotional well-being. It is well-validated, reliable, and responsive and will be administered to participants with COPD. Score range 0-6 with higher scores indicate worse health status.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 105 | 101
score on a scale | 3.08 (0.1) | 3.21 (0.1)

6. Secondary Outcome: Quality of Life at the End of Life (QUAL-EC)
Description: The QUAL-EC is a valid and reliable self-report measure of several domains, each scored separately, of quality of life in advanced illness. Each item is rated from 1 to 5, and mean scores for multiple items in a domain, i.e., subscale were estimated. Minimum score for each subscale is 1, maximum is 5. A higher score is a better perception of quality of life for each subscale.
Time Frame: 6 months
Population: Survey completeness differed by measure.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 154 | 152
score on a scale
  QUAL-E: Life Completion | 3.01 (0.23) | 2.88 (0.23)
  QUAL-E: Relationship With Healthcare Provider | 3.05 (0.22) | 2.87 (0.22)
  QUAL-E: Preparation | 3.86 (0.22) | 3.55 (0.22)
  QUAL-E: Feel At Peace: number analyzed (Participants) | 153 | 152
  QUAL-E: Feel At Peace | 3.35 (0.29) | 3.18 (0.29)

7. Secondary Outcome: Advance Care Planning Communication and Documentation
Description: Advance care planning discussions and advance directive documentation in the electronic medical record will be assessed via electronic medical record review. An advance directive includes either a living will and/or durable power of attorney for health care.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 154 | 152
Participants
  Documented Advance Care Planning Discussion | 106 | 5
  Documented Advance Directive | 58 | 62

8. Secondary Outcome: Mortality
Description: The following events will be assessed during the study period through medical record review to supplement patient report: mortality.
Time Frame: 12 months
Population: Number of deaths is reported
Measure: Number; unit: participants
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 154 | 152
participants | 6 | 5

9. Secondary Outcome: Generalized Anxiety Disorder Scale (GAD-7)
Description: The GAD-7 is a valid and reliable self-report measure of anxiety tested in medically ill outpatient populations. Score range 0-21 and higher scores indicate more anxiety symptoms.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 154 | 152
score on a scale | 5.82 (1.43) | 6.92 (1.42)

10. Secondary Outcome: Advance Care Planning Engagement
Description: This survey was designed to measure behaviors related to surrogate decision makers, values and quality of life, and informed decision making. Specifically, the Advance Care Planning-4 (ACP-4) measure (Sudore et al) was used.
  Minimum value is 1, maximum value is 5. Higher scores indicate higher levels of readiness to engage in advance care planning.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 154 | 152
score on a scale | 4.21 (0.34) | 3.68 (0.34)

11. Secondary Outcome: PEG (Pain)
Description: The PEG measures pain intensity and interference (Krebs, 2009). Scale range 0-10 and higher score indicates more pain.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 152 | 152
score on a scale | 4.76 (0.72) | 5.04 (0.72)

12. Secondary Outcome: Insomnia Severity Index (ISI)
Description: The ISI measures insomnia severity (Bastien, 2000). There are 6 items and a mean was used. Minimum score is 0, maximum score is 4. A higher score indicates more severe insomnia.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 153 | 152
score on a scale | 2.11 (0.26) | 2.26 (0.26)

13. Secondary Outcome: PROMIS Fatigue
Description: The Patient Reported Outcome Measurement Information System- Fatigue (PROMIS fatigue) measures fatigue severity. Scale range 0-4 and a higher score indicates more fatigue.
Time Frame: 6 months
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 153 | 152
score on a scale | 2.15 (0.26) | 2.22 (0.26)

14. Secondary Outcome: K-BILD
Description: Quality of life measure for interstitial lung disease. Score range 15-105 (lower score indicates lower health status).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 5 | 5
score on a scale | 54.8 (17.4) | 50.8 (5.8)

15. Secondary Outcome: Goal Concordance
Description: Two questions with Likert scale responses of 1 to 10: (1) Kind of medical care is most important to you; answers range from 0 = I prefer medical care that focuses on extending life, even if it means having more pain and discomfort, to 10 = I prefer medical care that focuses on relieving pain and discomfort, even if it means not living as long. (2) Medical care right now; answers range from 0 = My current medical care is focused on extending life, even if it means having more pain and discomfort to 10 = My current medical care is focused on relieving pain and discomfort, even if it means not living as long. Goal concordant = answers of 0-3 for both questions, 4-6 for both questions, or 7-10 for both questions. Patients who answered "I am not sure of the goals of my medical care" were considered "unsure of care focus."
Time Frame: 6 months
Population: Number analyzed = # of patients who we had complete data at 6 months and who were not unsure of their goals of care at the 6-month time point.
  The count of participants in the outcome measure data table is the number of patients who were considered goal concordant at 6 months for the control/intervention groups; this is the number of people who meet the criteria listed (Patients who answered 0-3 for both questions, 4-6 for both questions, or 7-10 for both questions).
Measure: Count of Participants; unit: Participants
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 85 | 85
Participants | 52 | 55

16. Secondary Outcome: Hospitalization
Description: The following events will be assessed during the study period through medical record review to supplement patient report: hospitalizations.
Time Frame: 6 months
Population: participants
Measure: Number; unit: participants
Arm/Group | ADAPT Intervention | Enhanced Usual Care
Number analyzed (Participants) | 154 | 152
participants
  Hospitalized Once | 24 | 17
  Hospitalized Twice or More | 9 | 9

ADVERSE EVENTS:
Time Frame: Adverse event reporting is reported from the time participants were randomized until 6-months (for hospitalizations and all other adverse events) and 12-months (for mortality).
Description: Serious adverse events included hospitalizations and mortality. Other adverse events (collected non-systematically) included events reported by patients or viewed in medical records. For example, ED visits, potential medication side effects, or symptoms of disease exacerbation/progression. Other adverse events were tracked more carefully (and more likely to be reported) in the intervention arm due to increased interventionist contact with participants compared to the enhanced usual care arm.
Arm/Group | ADAPT Intervention | Enhanced Usual Care
All-Cause Mortality (participants affected / at risk) | 6/154 | 5/152
Serious Adverse Events (participants affected / at risk) | 39/154 | 31/152
Other Adverse Events (participants affected / at risk) | 70/154 | 34/152
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADAPT Intervention (N=154) | Enhanced Usual Care (N=152)
Hospitalization (General disorders) | 33 | 26 — Hospitalizations were determined at 6 months and not adjudicated as to organ-specific cause.
Mortality (General disorders) | 6 | 5 — Mortality was determined at 1 year and was not adjudicated as to organ-specific cause.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ADAPT Intervention (N=154) | Enhanced Usual Care (N=152)
All other AEs (not SAE) (General disorders) | 70 | 34 — Anticipated and unanticipated events within any arm of the study were reported. AEs were more likely to be reported by intervention arm subjects due to more exposure to intervention staff. Hospitalizations, deaths, emergency room visits reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/47/NCT02713347/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-15): https://cdn.clinicaltrials.gov/large-docs/47/NCT02713347/SAP_001.pdf